CLINICAL TRIAL: NCT05981079
Title: Model-based Dose Versus Empirical Dose of Piperacillin/Tazobactam in the Treatment of Late-onset Sepsis in Preterm Neonates: a Multicentre, Randomised, Open-label, Non-inferiority Study.
Brief Title: Model-based Dose Versus Empirical Dose of Piperacillin/Tazobactam in Preterm Neonates With Late-onset Sepsis.
Acronym: PIP/TAZO
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shandong University (Other)
Collaborators: Shandong Provincial Hospital (Other Government); Qianfoshan Hospital (Other); Jinan Maternity and Child Care Hospital (Unknown); Yantai Yuhuangding Hospital (Other); Hebei Petro China Center Hospital (Unknown); Shengli Oilfield Hospital (Other); Liaocheng People's Hospital (Other); Jining Medical University (Other); W.F. Maternal and Child Health Hospital (Unknown); Taian City Central Hospital (Other)
Responsible Party: Principal Investigator, Wei Zhao, Head of department of clinical pharmacy and pharmacology, Shandong University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SDU-2023-NeoPIP-002
Record Dates: First submitted 2023-07-14; First posted 2023-08-08 (Actual); Last update posted 2023-08-08 (Actual); Status verified 2023-07

CONDITIONS: Late-Onset Neonatal Sepsis
Keywords: late-onset sepsis; piperacillin/tazobactam; model-based dose; empirical dose
MeSH Terms: conditions — Neonatal Sepsis | interventions — Piperacillin, Tazobactam Drug Combination

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Model-based dosing regimen (Experimental): Drug: Piperacillin Sodium and Tazobactam Sodium for Injection. Dosing regimen: GA<28 weeks: 30 mg/kg, Q8H; 28 weeks ≤GA<34 weeks: 50 mg/kg，Q8H.
  Interventions: Drug: Piperacillin/tazobactam
- Empirical dosing regimen (Active Comparator): Drug: Piperacillin Sodium and Tazobactam Sodium for Injection. Dosing regimen: 90 mg/kg，Q8H.
  Interventions: Drug: Piperacillin/tazobactam

INTERVENTIONS:
Drug: Piperacillin/tazobactam — Piperacillin Sodium and Tazobactam Sodium for Injection

SUMMARY:
This study aims to compare the clinical outcomes, safety and PD target attainment of the model-based dose and empirical dose of piperacillin/tazobactam in the treatment of LOS in premature neonates, so as to optimize the piperacillin/tazobactam dose regimen.

ELIGIBILITY:
Inclusion Criteria:

* Preterm neonates: gestational age <34 weeks;
* Postnatal age > 72h;
* Postmenstrual age <36 weeks;
* Newly diagnosed as late-onset sepsis;
* Parental written consent.

Exclusion Criteria:

* Patient with bacterial meningitis, osteomyelitis, septic arthritis or necrotizing enterocolitis requiring surgery.
* High suspicion of/confirmed fungal infection.
* Severe congenital malformations and/or severe organ failure.
* Administration of any systemic antibiotic regimen 24 h before screening.
* Administration of other systemic trial drug therapy.
* Other factors that the researcher considers unsuitable for inclusion.
* Post-randomization Exclusion: ①Patients with a positive baseline blood culture and the pathogen resistant to PIP/TAZO. ②Patients with bacterial meningitis, fungal infection, osteomyelitis, septic arthritis or necrotizing enterocolitis requiring surgery after randomization.

Min Age: 72 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 332 (Estimated)
Dates: Start 2023-07-31 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
Successful outcome | At the follow-up visit (10 ± 1 days after the end of actual piperacillin/tazobactam therapy )
  Successful outcome is defined as:
  1. Participant is alive.
  2. No need for replacing the antibiotic or adding new antibiotics.
  3. At the end of actual piperacillin/tazobactam therapy, ①there is a significant improvement in the participant's overall clinical status, ②there is microbiological resolution or presumed eradication of bacteria and ③no new piperacillin/tazobactam-susceptible pathogens potentially associated with sepsis have been identified.
  4. Participant does not have a clinically or microbiologically significant relapse or new infection within 10 days after the end of actual piperacillin/tazobactam therapy.

SECONDARY OUTCOMES:
Length of NICU stay | From the date of randomization until date of discharge, assessed up to 2 months
  Duration of hospital admission (days)
All cause in-hospital mortality | From the date of randomization until date of discharge, assessed up to 2 months
  Death before discharge from NICU
Proportion of patients switching to or adding another antibiotics. | Through study completion, an average of 20 days.
  Proportion of patients switching to or adding another antibiotics by any reason.
Relapsed or new infection rate | At the follow-up visit (10 ± 1 days after the end of actual piperacillin/tazobactam therapy )
  Proportion of patients with clinically or microbiologically significant relapsed or new infection.
PD target attainment | Through study completion, an average of 20 days.
  70%fT>MIC
Adverse events | Through study completion, an average of 20 days.
  Drug-related adverse events and serious adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Wei Zhao, Ph.D, Principal Investigator — Shandong University
Locations (10):
- China (10):
  - Shengli Oilfield Hospital, Dongying
  - Jinan Maternity and Child Care Hospital, Jinan
  - Qianfoshan Hospital, Jinan
  - Shandong Provincial Hospital, Jinan
  - Jining Medical University, Jining
  - Hebei Petro China Center Hospital, Langfang
  - Liaocheng People's Hospital, Liaocheng
  - Taian City Central Hospital, Tai’an
  - W.F. Maternal and Child Health Hospital, Weifang
  - Yantai Yuhuangding Hospital, Yantai